CLINICAL TRIAL: NCT01142869
Title: An Observational Study to Evaluate the Safety and Efficacy of Cetuximab in Combination With Platinum-based Chemotherapy, in the First-line Therapy of Recurrent/ Metastatic Squamous Cell Carcinoma of Head and Neck (SCCHN)
Brief Title: An Observational Study to Evaluate the Safety and Efficacy of Cetuximab in Combination With Platinum-based Chemotherapy in the First-line Treatment of Recurrent or Metastatic Squamous Cell Carcinoma of Head and Neck
Status: Terminated | Type: Observational
Why Stopped: The study was discontinued due to slow recruitment and subjects not completing follow up period.
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Ltd., India (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR 062202-514
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Carcinoma, Squamous Cell
Keywords: Carcinoma, Squamous Cell; Erbitux; Neoplasms, Squamous Cell
MeSH Terms: conditions — Carcinoma, Squamous Cell; Neoplasms, Squamous Cell | interventions — Cetuximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood

INTERVENTIONS:
Drug: Cetuximab — The starting dose will be intravenous (IV) cetuximab 400 mg/m2 body surface area administered as a 120-minute infusion once a week . The subsequent weekly doses will be IV cetuximab 250 mg/m2 administered as a 60-minute infusion. The maximum infusion rate must not exceed 10 mg/min.
  Other Names: Erbitux

SUMMARY:
The aim of this prospective, observational, multicenter, post-marketing study is to evaluate the safety and efficacy of Cetuximab (Erbitux) in combination with platinum based chemotherapy, in the first line therapy of recurrent/ metastatic squamous cell carcinoma of head and neck (SCCHN). A total of 100 subjects with SCCHN will be recruited in 20 centres across India.

ELIGIBILITY:
Inclusion Criteria:

* The study inclusion criteria is as per the label for patients with metastatic/recurrent SCCHN approved by India Health Authorities, i.e., "Cetuximab is indicated for the treatment of patients with squamous cell cancer of the head and neck in combination with platinum-based chemotherapy for recurrent and/or metastatic disease."
* For each platinum-based chemotherapy, the related product labels approved by India Health Authorities will also be followed strictly in terms of patient eligibility.

Exclusion Criteria:

* Patients with known severe (grade 3 or 4; National Cancer Institute-Common Toxicity Criteria [NCI-CTC]) hypersensitivity reactions to Cetuximab are contraindicated for Cetuximab

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with squamous cell carcinoma of head and neck
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2009-12-31 (Actual); Primary Completion 2013-07-31 (Actual); Study Completion 2014-08-05 (Actual)

PRIMARY OUTCOMES:
To obtain further safety information on the use of Cetuximab in combination with platinum-based chemotherapy in patients with recurrent/metastatic SCCHN. | From first infusion of cetuximab until 28 days after the last infusion.
  Safety variables will include the assessment of incidence and type of adverse drug reactions (ADRs), serious adverse drug reactions (SADRs), incidence of withdrawals due to intolerability of cetuximab and severity of adverse events (AEs)

SECONDARY OUTCOMES:
To obtain clinical effectiveness information of Cetuximab in combination with platinum based chemotherapy in patients with recurrent/ metastatic SCCHN. | From first infusion of cetuximab until 28 days after the last infusion.
  Clinical efficacy will be assessed by best tumor response, disease control rate, progression-free survival and overall survival with cetuximab treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Rajiv Rana, Study Director — Merck Ltd., India
Locations (28):
- India (28):
  - Ambaa Hospitals, Hyderabad, Andhra Pradesh
  - Indo- American Cancer Institute & Research Centre, Hyderabad, Andhra Pradesh
  - NVS Ramakrishna's Clinic, Hyderabad, Andhra Pradesh
  - Dr. Nikhil's Clinic, Secunderabad, Andhra Pradesh
  - Swarna Sai Hospital, Secunderabad, Andhra Pradesh
  - Sparsh Hospital, Orissa, Bhubaneswar
  - Wellness Consultants Clinic, Surat, Gujarat
  - Global Health Pvt Ltd, Gurgaon, Haryana
  - The Cancer Clinic, Kochi, Kerala
  - Dr. T. P. Sahoo's Clinic, Bhopal, Madhya Pradesh
  - BND Onco Centre, Mumbai, Maharashtra
  - S.L.Raheja Hospital, Mumbai, Maharashtra
  - S M Karandikar's Clinic, Pune, Maharashtra
  - Ruby Hall Clinic, Pune, Maharashtra
  - Galaxy Care Laproscopic Institute, Pune, Maharashtra
  - Neigrihms, Shillong, Meghālaya
  - Grace Nursing Home, Aizawl, Mizoram
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Cancer Clinic, Jaipur, Rajasthan
  - SMS Hospital, Jaipur, Rajasthan
  - Bhagwan Mahaveer Cancer Hospital, Jaipur, Rajasthan
  - J.K.Cancer Institute, Kanpur, Uttar Pradesh
  - Annapurna Medical and Cancer Relief Society, Lucknow, Uttar Pradesh
  - Dr. Vineet's Clinic, New Delhi, Uttar Pradesh
  - SMH-Curie Cancer Centre, Shanti Mukand Hospital, New Delhi, Uttar Pradesh
  - B.R. Singh Hospital, Kolkata, West Bengal
  - Apollo Gleneagles Cancer Hospital, Kolkata, West Bengal
  - Sunil Gupta's Clinic, Delhi